CLINICAL TRIAL: NCT05704322
Title: The Effectiveness of the Wim Hof Method on Physical and Mental Health of People with a Spinal Cord Injury
Brief Title: The Effectiveness of the Wim Hof Method in People with Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting Reade (Other)
Collaborators: Dr. C.J. Vaillant Fonds (Unknown); W.M. de Hoop Stichting (Unknown); Ars Donandi / Yske Walther fonds (Unknown); Reade foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W22.069; NL81525.015.22 (Other: CCMO)
Record Dates: First submitted 2022-12-29; First posted 2023-01-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual care group (No Intervention): The control group will not receive any intervention, they will receive usual care and only participate in the pre and post tests.
- Wim Hof Method - breathing and mindset exercise (Experimental): The first intervention group will practice the breathing and mindset exercise.
  Interventions: Other: Wim Hof Methode
- Wim Hof Method - breathing and mindset exercise and cold exposure (Experimental): The second intervention group will also practice the cold exposure (i.e, breathing, mindset and cold exposure)
  Interventions: Other: Wim Hof Methode

INTERVENTIONS:
Other: Wim Hof Methode — The intervention groups will follow a 7-weeks intervention, with one practice session per week at the rehabilitation center led by Wim Hof or one of his instructors. Besides these joint weekly sessions, the intervention groups have to practice daily at home with the Wim Hof Method app.
  Arms: Wim Hof Method - breathing and mindset exercise; Wim Hof Method - breathing and mindset exercise and cold exposure

SUMMARY:
People with a spinal cord injury (SCI) often experience secondary medical complications. One of the methods that may help to prevent or deal with secondary complications in people with SCI is the Wim Hof Method (WHM). The WHM is based on three elements: 1) breathing exercises, 2) gradual cold exposure (cold showers, or cold water immersion), and 3) mindset. The primary objective of this randomized controlled trial is to assess the effects of WHM, involving breathing exercises, mindset (and cold exposure), on health-related quality of life in people with SCI. The secondary objectives are to assess the effects of WHM, involving breathing exercises, mindset (and cold exposure) in people with SCI on: inflammation markers, metabolic health, pulmonary function, body composition, sleep quality, spasticity, stress, and on chronic pain.

DETAILED DESCRIPTION:
A spinal cord injury (SCI) is a serious medical condition that causes functional, psychological and socioeconomic disorder. Long-term, secondary medical complications are common and play an important role in the continuum of care for people with SCI. Complications are a frequent cause of morbidity and mortality and lead to increased rates of rehospitalisation, loss of employability and decreased quality of life. During multidisciplinary SCI rehabilitation, the treatment is focussed on working with the patient physically and psychologically to maximize their neurological recovery and general health but also to prevent or deal with the secondary complications. One of the methods that may help to prevent or deal with secondary complications in people with SCI is the Wim Hof Method (WHM). The WHM is based on three elements: 1) breathing exercises, 2) gradual cold exposure (cold showers, or cold water immersion), and 3) mindset. Previous studies showed a positive effect of the WHM on health-related quality of life and the inflammatory profile of healthy individuals as well as patients with active axial spondyloarthritis. Furthermore, a pilot study in people with SCI showed that the WHM (only breathing exercises and mindset) led to positive changes in respiratory function, mental health index, hyperventilation and a trend was visible regarding the hindrance due to spasticity. Some of the participants mentioned that they experienced positive effects on coughing, energy level, mood or used less spasticity medication after the WHM intervention. These positive findings in the pilot study warrant a full-scale randomised-controlled trial (RCT) of this novel therapeutic approach in people with SCI.

The primary objective of this randomized controlled trial is to assess the effects of WHM, involving breathing exercises, mindset (and cold exposure), on health-related quality of life in people with SCI. The secondary objectives are to assess the effects of WHM, involving breathing exercises, mindset (and cold exposure) in people with SCI on: inflammation markers, metabolic health, pulmonary function, body composition, sleep quality, spasticity, stress, and on chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (Male/Female) with either a complete or incomplete chronic SCI. In this study, a chronic SCI is defined as a time since injury ≥ 1 year.
* Participants have to be between 18 and 75 years old.

Exclusion Criteria:

* Cardiac arrhythmias or cardiac disease;
* A history of severe autonomic dysreflexia assessed with the 'Autonomic standards assessment';
* Severe pulmonary disease (such as COPD) based on a pulmonary history;
* Insufficient mastery of the Dutch language (speaking and reading);
* Severe cognitive or communicative disorders;
* Progressive disease;
* Being or becoming pregnant during the study period;
* Severe psychiatric illness or disorders (at the discretion of the treating rehabilitation physician);
* Involved in another intervention study which may have an effect on the outcome measures of the present study;
* Experience with (parts of) the Wim Hof Method.
* Negative advice from physician to participate in the Wim Hof Method intervention based on the medical screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in mental health | Assessed before and after the 7-weeks WHM intervention
  Mental Health Index - 5 (MHI-5), a subscale of the SF-36. The MHI-5 has a score of 0 to 100, where a score of 100 represents optimal mental health.

SECONDARY OUTCOMES:
Change in health-related quality of life | Assessed before and after the 7-weeks WHM intervention
  The SF-36 measures measures eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each scale is scored on a 0 to 100 range, a higher score defines a more favorable health state.
Change in mindful attention awareness | Assessed before and after the 7-weeks WHM intervention
  The Mindful Attention Awareness Scale is a 15-item scale designed to assess a core characteristic of mindfulness. Each item can be scored from 1 (almost always) to 6 (almost never). The overall outcome is the average of the 15 items, with a higher score indicating being more mindful.
Change in hyperventilation | Assessed before and after the 7-weeks WHM intervention
  The Nijmegen Hyperventilation Syndrome Questionnaire has 16 items (related to symptoms of hyperventilation syndrome) to be answered on a 5-point scale ranging from 'never' (0) to 'very often' (4). A total score of more than 23 out of 64 points suggests significant hyperventilation.
Change in pain and pain interference | Assessed before and after the 7-weeks WHM intervention
  Four questions of the International Spinal Cord Injury Pain basic data set will be used to assess (the interference of) pain on a 0 (no pain or no interference) to 10 (extreme pain or extreme interference) range.
Change in sleep quality | Assessed before and after the 7-weeks WHM intervention
  Pittsburgh Sleep Quality Index (PSQI) is a self-rating questionnaire resulting in a global score between 0 and 21, which consists of seven subscores. Higher scores indicate worse sleep quality.
Change in hindrance due to spasticity | Assessed before and after the 7-weeks WHM intervention
  Hindrance due to spasticity will be assessed with a subjective rating scale for each of the following activities: (1) sleeping; (2) making transfers; (3) washing and clothing; (4) wheelchair driving; (5) 'others'. The scale ranges from 0 to 2 (0: no hindrance due to spasticity; 1: little hindrance due to spasticity; 2: a lot of hindrance due to spasticity). A sum score for hindrance during all activities will be calculated. It ranges from 0 (no hindrance) to 10 (a lot of hindrance during all activities).
Change in CRP | Assessed before and after the 7-weeks WHM intervention
  Concentration CRP (mg/L) in blood
Change in IL-6 | Assessed before and after the 7-weeks WHM intervention
  Concentration IL-6 (pg/ml) in blood
Change in fasted glucose | Assessed before and after the 7-weeks WHM intervention
  Concentration of fasted glucose (mmol/l) in blood
Change in triglycerides | Assessed before and after the 7-weeks WHM intervention
  Concentration of triglycerides (mmol/l) in blood
Change in high-density lipoprotein | Assessed before and after the 7-weeks WHM intervention
  Concentration of high-density lipoprotein (mmol/l) in blood
Change in low-density lipoprotein | Assessed before and after the 7-weeks WHM intervention
  Concentration of low-density lipoprotein (mmol/l) in blood
Change in total cholesterol | Assessed before and after the 7-weeks WHM intervention
  Concentration of total cholesterol (mmol/l) in blood
Change in blood pressure | Assessed before and after the 7-weeks WHM intervention
  Systolic and diastolic blood pressure (mm Hg)
Change in forced vital capacity | Assessed before and after the 7-weeks WHM intervention
  Forced vital capacity (FVC, liter) measured by spirometry
Change in forced expiratory volume | Assessed before and after the 7-weeks WHM intervention
  Forced expiratory volume in 1 sec (FEV1, liter) measured by spirometry
Change in forced inspiratory volume | Assessed before and after the 7-weeks WHM intervention
  Forced inspiratory volume in 1 sec (FIV1, liter) measured by spirometry
Change in peak expiratory flow | Assessed before and after the 7-weeks WHM intervention
  Peak expiratory flow (PEF, liter/s) measured by spirometry
Change in peak inspiratory flow | Assessed before and after the 7-weeks WHM intervention
  Peak inspiratory flow (PIF, liter/s) measured by spirometry
Change in body mass | Assessed before and after the 7-weeks WHM intervention
  Body mass (kg) measured on a (wheelchair) weighing scale
Change in fat and fat free mass | Assessed before and after the 7-weeks WHM intervention
  Fat mass and fat free mass (both in kg) measured by bio-impedance analysis:
Participant compliance and experiences | Assessed before and after the 7-weeks WHM intervention
  Diary and exit interview

CONTACTS AND LOCATIONS:
Overall Officials: Sonja de Groot, PhD, Principal Investigator — Stichting Reade
Locations (1):
- Stichting Reade, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoekstra S, Ettema F, van der Bijll M, van der Sterren V, van Binsbergen E, van Orsouw L, Achterberg W, Daanen H, Janssen T, de Groot S. The effect of breathing exercises and mindset with or without cold exposure on mental and physical health in persons with a spinal cord injury-a protocol for a three-arm randomised-controlled trial. Spinal Cord. 2024 May;62(5):237-240. doi: 10.1038/s41393-024-00976-9. Epub 2024 Mar 15. PMID 38491303